CLINICAL TRIAL: NCT04186572
Title: Usefulness of the Variation of the CLIF-C ACLF Score in Patients With Acute on Chronic Liver Failure
Acronym: ARIHAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Nestor Pistillo, Head of Intensive Care Unit at Hospital El Cruce, Hospital El Cruce
Other Study IDs: HCruce
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: Acute-On-Chronic Liver Failure; Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Liver Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with Acute on Chronic Liver Failure (ACLF) have high short-term mortality. The use of a severity score could define the patient's prognosis and would help determine in whom the treatment is effective or futile.

DETAILED DESCRIPTION:
Acute on Chronic Liver Failure (ACLF) is a syndrome characterized by the presence of an acute decompensation of cirrhosis, associated with failure of at least one other organ or extra hepatic system. It is characterized by high mortality in the short term and its prevalence varies between countries and regions.

It is an extraordinarily dynamic entity in which more than 50% of patients with less severe forms improve, while in those with 3 or more organ failures, the transplant rate is low and mortality is 90%. It is important to highlight that those patients with ACLF who manage to be transplanted have the same survival as cirrhotic patients without ACLF. There is no specific treatment, only life support and early determination of the precipitating factor and its eventual resolution.

Having tools that define the short-term prognosis of these patients, especially the variation of the score (CLIF-C ACLF) during the first week, would have an important clinical relevance, because it can help define the patients who benefit from the supportive treatment and in whom the therapeutic effort is futile.

The biomarker Neutrophil Gelatinase-Associated Lipocalin (NGAL) is increased in plasma and urine in patients with ACLF and could help improve the prognostic ability of the CLIF-C ACLF score.

ELIGIBILITY:
Inclusion Criteria:

* Acute on Chronic Liver Failure

Exclusion Criteria:

* Acute liver failure, terminal disease, pregnancy, previous liver transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis with ACLF over 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the degree of severity of the ACLF with the CLIF-C ACLF score at the time of diagnosis and its variation on day 3 and 7 | one week
  The severity of the ACLF will be assessed by means of a score (CLIF_C ACLF) at the time of admission, day three and seven. Good evolution of the score will be considered when it decreases and bad evolution when it remains the same or increases.

SECONDARY OUTCOMES:
Correlate the variation of the score (CLIF-C ACLF) and mortality at 28, 60 and 90 days. | 90 days
  The variation of the score (good or bad evolution) will be correlated with mortality at 28, 60 and 90 days.
ACLF epidemiological evaluation. | 90 days
  Incidence, prevalence of ACLF will be determined. Triggers (hepatic and / or extra hepatic causes).
Correlate the level of NGAL with the development of ACLF and its severity evaluated by the CLIF-C ACLF score. | 1 day
  The level of NGAL in plasma and urine will be determined routinely at the time of diagnosis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreau R, Jalan R, Gines P, Pavesi M, Angeli P, Cordoba J, Durand F, Gustot T, Saliba F, Domenicali M, Gerbes A, Wendon J, Alessandria C, Laleman W, Zeuzem S, Trebicka J, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Acute-on-chronic liver failure is a distinct syndrome that develops in patients with acute decompensation of cirrhosis. Gastroenterology. 2013 Jun;144(7):1426-37, 1437.e1-9. doi: 10.1053/j.gastro.2013.02.042. Epub 2013 Mar 6. PMID 23474284
- [Background] Jalan R, Gines P, Olson JC, Mookerjee RP, Moreau R, Garcia-Tsao G, Arroyo V, Kamath PS. Acute-on chronic liver failure. J Hepatol. 2012 Dec;57(6):1336-48. doi: 10.1016/j.jhep.2012.06.026. Epub 2012 Jun 28. PMID 22750750
- [Background] Gustot T, Fernandez J, Garcia E, Morando F, Caraceni P, Alessandria C, Laleman W, Trebicka J, Elkrief L, Hopf C, Solis-Munoz P, Saliba F, Zeuzem S, Albillos A, Benten D, Montero-Alvarez JL, Chivas MT, Concepcion M, Cordoba J, McCormick A, Stauber R, Vogel W, de Gottardi A, Welzel TM, Domenicali M, Risso A, Wendon J, Deulofeu C, Angeli P, Durand F, Pavesi M, Gerbes A, Jalan R, Moreau R, Gines P, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Clinical Course of acute-on-chronic liver failure syndrome and effects on prognosis. Hepatology. 2015 Jul;62(1):243-52. doi: 10.1002/hep.27849. Epub 2015 May 29. PMID 25877702
- [Background] Bajaj JS, O'Leary JG, Reddy KR, Wong F, Biggins SW, Patton H, Fallon MB, Garcia-Tsao G, Maliakkal B, Malik R, Subramanian RM, Thacker LR, Kamath PS; North American Consortium For The Study Of End-Stage Liver Disease (NACSELD). Survival in infection-related acute-on-chronic liver failure is defined by extrahepatic organ failures. Hepatology. 2014 Jul;60(1):250-6. doi: 10.1002/hep.27077. Epub 2014 May 29. PMID 24677131